CLINICAL TRIAL: NCT02950766
Title: A Phase I Study Combining NeoVax, a Personalized NeoAntigen Cancer Vaccine, With Ipilimumab to Treat High-risk Renal Cell Carcinoma
Brief Title: NeoVax Plus Ipilimumab in Renal Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Patrick Ott, MD, PhD (Other)
Collaborators: Bristol-Myers Squibb (Industry); Oncovir, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Patrick Ott, MD, PhD, MD, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-097
Record Dates: First submitted 2016-09-08; First posted 2016-11-01 (Estimated); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Kidney Cancer
Keywords: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Neovax in Combination with Ipilimumab (Experimental): Patients will undergo surgery with the intent to resect the primary kidney tumor
  Neovax is a combination of Poly-ICLC and Neoantigen Peptides
  Priming doses of NeoVax will be administered on days 1, 4, 8, 15, and 22
  * In the boost phase, vaccine will be administered on days 78 (week 12) and 134 (week 20
  Ipilimumab will be injected within 1 cm of each NeoVax administration
  Interventions: Drug: NeoVax; Drug: Ipilimumab
- NeoVax alone (Experimental): Patients will undergo surgery with the intent to resect the primary kidney tumor
  Neovax is a combination of Poly-ICLC and Neoantigen Peptides
  Priming doses of NeoVax will be administered on days 1, 4, 8, 15, and 22
  * In the boost phase, vaccine will be administered on days 78 (week 12) and 134 (week 20)
  Interventions: Drug: NeoVax

INTERVENTIONS:
Drug: NeoVax — combination of Neoantigen peptides and poly-ICLC
  Other Names: neoantigen vaccine
Drug: Ipilimumab — local administration of ipilimumab
  Other Names: Yervoy
  Arms: Neovax in Combination with Ipilimumab

SUMMARY:
This research study is evaluating a new type of Kidney Cancer vaccine called "Personalized NeoAntigen Cancer Vaccine"as a possible treatment for Kidney Cancer.

The following intervention will be involved in this study:

* Personalized Neoantigen Vaccine
* Poly-ICLC (Hiltonol)
* Ipilimumab

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational kidney cancer vaccine and also tries to define the appropriate dose of the investigational kidney cancer vaccine to use for further studies. "Investigational" means that the kidney cancer vaccine, in this case the Personalized Neoantigen Cancer Vaccine, is being studied. It also means that the FDA (the U.S. Food and Drug Administration) has not approved the Personalized Cancer Vaccine for any use in patients, including people with kidney cancer.

Poly-ICLC (also called Hiltonol) is an experimental "viral mimic" and an activator of immunity. Poly-ICLC is an investigational drug, meaning the FDA has not approved it as a treatment for any disease.

Personalized NeoAntigen Cancer Vaccine: The purpose of this study is to determine if it is possible to make and administer safely a vaccine against kidney cancer by using information gained from specific characteristics of the participant's own kidney cancer. It is known that kidney cancers have mutations (changes in genetic material) that are specific to an individual patient and tumor. These mutations can cause the tumor cells to produce proteins that appear very different from the body's own cells. It is possible that these proteins used in a vaccine may induce strong immune responses, which may help the participant's body fight any tumor cells that could cause the kidney cancer to come back in the future. The study will examine the safety of the vaccine when given at several different time points and will examine the participant's blood cells for signs that the vaccine induced an immune response.

Ipilimumab (Yervoy™) is an antibody that has been approved by the United States Food and Drug Administration (FDA) for the treatment of melanoma.

In this research study, the investigators are looking at the safety and tolerability of the Personalized NeoAntigen Cancer Vaccine combined with Ipilimumab as well as the body's immune response to the vaccine. Ipilimumab will be delivered as an injection given underneath the skin rather than injected in the vein in proximity to each vaccination site in order to 1) direct anti-CTLA4 activity to the vaccine-draining lymph nodes and 2) limit potential toxic effects.

ELIGIBILITY:
Inclusion Criteria for Initial Registration:

* Ability to understand and the willingness to sign a written informed consent document.
* Patients should have suspected stage III or stage IV clear cell renal cell carcinoma (ccRCC), with anticipation that all disease can be surgically resected. Confirmation of clear cell histology, final stage (III or IV), and removal of all disease will be done after the surgery, and will be required for further participation of the trial.
* Patient is agreeable to allow tumor and normal tissue samples to be submitted for complete exome and transcription sequencing.
* Patients undergoing a potentially curative metastatectomy are eligible if the tumor tissue from the surgery is enough to make a vaccine.
* ECOG (Eastern Cooperative Oncology Group) performance status ≤ 1.
* Age ≥ 18 years.
* Participants must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL (microliter)
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * AST (SGOT) /ALT (SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine clearance ≥40 mL/min/(calculated using the Cockroft-Gault equation)
* Women of childbearing potential (WOCBP) must have a negative pregnancy test (minimum sensitivity 25 IU/L or equivalent of HCG) before entry onto the trial and within 7 days prior to start of study medication, because the effects NeoVax on the developing human fetus are unknown. It is the investigators' responsibility to repeat the pregnancy test should start of treatment be delayed.
* Female patients enrolled in the study, who are not free from menses for >2 years, post hysterectomy / oophorectomy, or surgically sterilized, must be willing to use either 2 adequate barrier methods or a barrier method plus a hormonal method of contraception to prevent pregnancy or to abstain from sexual activity for the duration of treatment with ipilimumab plus 5 half-lives of ipilimumab (75 days) plus 30 days (duration of ovulatory cycle) for a total of 105 days post-treatment completion. Approved contraceptive methods include for example: intra uterine device, diaphragm with spermicide, cervical cap with spermicide, male condoms, or female condom with spermicide. Spermicides alone are not an acceptable method of contraception.
* Male patients must agree to use an adequate method of contraception for the duration of treatment with study drugs plus 5 half-lives of the study drug (75 days) plus 90 days (duration of sperm turnover) for a total of 165 days post-treatment.

Eligibility Criteria for Secondary Registration

* ECOG performance status ≤1.
* Participants must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine ≥40 mL/min/(calculated using the Cockroft-Gault equation)
* Patients must have histologically confirmed clear cell renal cell carcinoma (ccRCC), stage III or fully resected stage IV (no evidence of disease), before starting study drugs per AJCC 8th edition.
* No evidence of disease (NED) at secondary registration.
* Women of childbearing potential (WOCBP) must have a negative pregnancy test (minimum sensitivity 25 IU/L or equivalent of HCG) within 7 days prior to start of study medication, because the effects NeoVax on the developing human fetus are unknown. It is the investigators' responsibility to repeat the pregnancy test should start of treatment be delayed.
* Female patients enrolled in the study, who are not free from menses for >2 years, post hysterectomy / oophorectomy, or surgically sterilized, must be willing to use either 2 adequate barrier methods or a barrier method plus a hormonal method of contraception to prevent pregnancy or to abstain from sexual activity throughout the study, starting with visit 1 through 4 weeks after the last dose of study therapy. Approved contraceptive methods include for example; intra uterine device, diaphragm with spermicide, cervical cap with spermicide, male condoms, or female condom with spermicide. Spermicides alone are not an acceptable method of contraception.
* Male patients must agree to use an adequate method of contraception for the duration of treatment with study drugs plus 5 half-lives of the study drug (75 days) plus 90 days (duration of sperm turnover) for a total of 165 days post-treatment.

Exclusion Criteria:

* Prior treatment with immune-modulatory agents including, but not limited to: IL-2, CTLA-4 blockade, PD-1/PD-L1 blockade, CD40 stimulation, or CD137 stimulation.
* Prior investigational ccRCC-directed cancer vaccine therapy.
* Patients with active brain metastases or leptomeningeal disease.
* Prior systemic therapy, including targeted therapy such as VEGF or mTOR inhibitors unless it is >6 months between last dose of drug and first vaccination with NeoVax. Systemic therapy is allowed only if prior therapy was not immune therapy (i.e. VEGF TKI), and it was >6 months ago.
* Treatment with other investigational products within the last 2 months prior to entry into this study.
* Previous bone marrow or stem cell transplant.
* Concomitant therapy with any anti-cancer agents for ACTIVE cancer treatment, other investigational anti-cancer therapies, or immunosuppressive agents; chronic use of systemic corticosteroids with prednisone >10 mg/day.
* Use of a non-oncology vaccine therapy for prevention of infectious diseases (with the exception of vaccination against the SARS-CoV-2 virus for the prevention of COVID-19 disease) is not allowed for 4 weeks prior to day 1, until 8 weeks after last study dose. Given the severity of the COVID-19 pandemic, vaccination specifically against the SARS-CoV-2 virus for the prevention of COVID-19 is ALLOWED in this study.
* History of severe allergic reactions attributed to any vaccine therapy for the prevention of infectious diseases.
* History of or current active autoimmune diseases, [e.g. including but not limited to inflammatory bowel diseases [IBD], rheumatoid arthritis, autoimmune thyroiditis, autoimmune hepatitis, systemic sclerosis (scleroderma and variants), systemic lupus erythematosus, autoimmune vasculitis, autoimmune neuropathies (such as Guillain-Barre syndrome). Vitiligo and adequately controlled endocrine deficiencies such as hypothyroidism are not exclusionary.].
* Patients who have had a history of acute diverticulitis, intra-abdominal abscess, GI obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation.
* Concomitant treatment with corticosteroids greater than physiologic doses (used in the management of cancer or non-cancer-related illnesses). Topical (if not including the proposed vaccination sites) or inhalational steroids are allowed.
* Known chronic infections with HIV, hepatitis B or C.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia.
* History of current immunodeficiency disease [e.g., splenectomy or splenic irradiation].
* Any underlying medical condition, psychiatric condition or social situation that in the opinion of the investigator would compromise study administration as per protocol or compromise the assessment of AEs.
* Pregnant women are excluded from this study because personalized neoantigen peptides and poly-ICLC are agents with unknown risks to the developing fetus. Because there is an unknown but potential risk of adverse events in nursing enfants secondary to treatment of the mother with personalized neoantigen peptides and poly-ICLC, nursing women are excluded from this study.
* Individuals with a history of another invasive malignancy are ineligible except for the following circumstances: a) individuals with a history of invasive malignancy are eligible if they have been disease-free for at least 2 years and are deemed by the investigator to be at low risk for recurrence of that malignancy; b) individuals with any of the following cancers are eligible if diagnosed and treated: carcinoma in situ of the breast, oral cavity or cervix and basal cell or squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2019-03-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicity (DLT) experienced within 49 days (7 weeks) of treatment initiation as assessed by CTCAE v4.0 | 49 days

SECONDARY OUTCOMES:
Number of participants with NeoVax induced IFN γ (interferon γ) T-cell Response against neoepitopes measured by ELISPOT at week 16 | 16 weeks
Number of participants alive at 2 years | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Ott, MD, Principal Investigator — Dana-Farber Cancer Institute; Toni Choueiri, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Braun DA, Moranzoni G, Chea V, McGregor BA, Blass E, Tu CR, Vanasse AP, Forman C, Forman J, Afeyan AB, Schindler NR, Liu Y, Li S, Southard J, Chang SL, Hirsch MS, LeBoeuf NR, Olive O, Mehndiratta A, Greenslade H, Shetty K, Klaeger S, Sarkizova S, Pedersen CB, Mossanen M, Carulli I, Tarren A, Duke-Cohan J, Howard AA, Iorgulescu JB, Shim B, Simon JM, Signoretti S, Aster JC, Elagina L, Carr SA, Leshchiner I, Getz G, Gabriel S, Hacohen N, Olsen LR, Oliveira G, Neuberg DS, Livak KJ, Shukla SA, Fritsch EF, Wu CJ, Keskin DB, Ott PA, Choueiri TK. A neoantigen vaccine generates antitumour immunity in renal cell carcinoma. Nature. 2025 Mar;639(8054):474-482. doi: 10.1038/s41586-024-08507-5. Epub 2025 Feb 5. PMID 39910301